CLINICAL TRIAL: NCT05808036
Title: The Efficacy of the DOMINO Diet Application Versus the Low FODMAP Diet in Tertiary Care IBS Patients
Brief Title: Efficacy of the DOMINO Diet App in IBS
Acronym: EDDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S67508
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: DOMINO; Low FODMAP diet; Irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: All patients will start with the DOMINO diet. Depending on the symptom improvement they will continue the DOMINO diet or switch to the strict low FODMAP diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DOMINO app - DOMINO app (Other): The patients start with the DOMINO diet (8 weeks). Patients that experienced symptom improvement, will continue with the DOMINO diet (6 weeks).
  Interventions: Other: Dietary intervention: DOMINO app
- DOMINO app - low FODMAP diet (Active Comparator): The patients start with the DOMINO diet (8 weeks). Patients that experienced no symptom improvement, will switch to the strict low FODMAP diet (6 weeks).
  Interventions: Other: Dietary intervention: DOMINO app; Other: Dietary intervention: low FODMAP diet

INTERVENTIONS:
Other: Dietary intervention: DOMINO app — Life style intervention and diet low in FODMAPs.
Other: Dietary intervention: low FODMAP diet — Strict low FODMAP diet.
  Arms: DOMINO app - low FODMAP diet

SUMMARY:
The aim of this study is to evaluate whether the DOMINO diet application is an effective tool in the treatment of Irritable bowel syndrome in tertiary care. Furthermore, this study aims to determine the response rate of the strict low FODMAP diet in non-responders to the DOMINO diet.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
3. Patients with irritable bowel syndrome according to Rome IV diagnostic criteria
4. Patients ages between 18 and 70 years old

Exclusion Criteria:

1. Participant has a history of any major psychiatric disorders (including those with a major psychosomatic element to their gastrointestinal disease), depression, alcohol or substance abuse in the last 2 years
2. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
3. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial
4. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive
5. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
6. Patients presenting with predominant symptoms of functional dyspepsia (FD) and of gastro-oesophageal reflux disease (GERD)
7. Patients following a diet interfering with the study diet in opinion of the investigator
8. Patients who already followed the low FODMAP diet under guidance of a trained dietitian without success

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-03 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Symptom response DOMINO app and low FODMAP diet | 18 months
  The symptom response is measured by the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS). In this questionnaire, each question (5) is scored from 0-100, with a maximum total score of 500. Improvement is defined as a 50-point or more drop on the IBS-SSS. The score is positively correlated with severity of IBS symptoms, a score from 50-175 indicated mild disease, 175-300 moderate and >300 severe.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No